CLINICAL TRIAL: NCT04664075
Title: Predicting Severity and Disease Progression in Influenza-like Illness
Brief Title: Predicting Severity and Disease Progression in Influenza-like Illness (Including COVID-19)
Acronym: PREDICT-ILI
Status: Terminated | Type: Observational
Why Stopped: The study failed to recruit sufficient number of participants.
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20SM6170
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Influenza; SARS (Severe Acute Respiratory Syndrome); Respiratory Viral Infection; Respiratory Tract Infections; Infection, Bacterial; Infection Viral; Covid19; RNA Virus Infections
Keywords: Flu; Influenza; SARS-CoV-2; Covid19; Respiratory; Predict; Infection; RNA
MeSH Terms: conditions — Influenza, Human; Severe Acute Respiratory Syndrome; Respiratory Tract Infections; Bacterial Infections; Virus Diseases; COVID-19; RNA Virus Infections; Infections | interventions — Cold Temperature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and nasal scrapes (using RhinoPro) for analysis by transcriptomics and qPCR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Respiratory infections — With biological samples and longitudinal observations, the aim is to find and develop predictive tests to better understand how and when flu-like illness progresses to more severe disease. This may help to decide which people need to be admitted to hospital, and how their treatment needs to be increased or decreased during infection.

SUMMARY:
Respiratory infections such as colds, flu and pneumonia affect millions of people around the world every year. Most cases are mild, but some people become very unwell. Influenza ('flu') is one of the most common causes of lung infection. Seasonal flu affects between 10% and 46% of the population each year and causes around 12 deaths in every 100,000 people infected. In addition, both influenza and coronaviruses have caused pandemics in recent years, leading to severe disease in many people. Although flu vaccines are available, these need to change every year to overcome rapid changes in the virus and are not completely protective.

This study aims to find and develop predictive tests to better understand how and when flu-like illness progresses to more severe disease. This may help to decide which people need to be admitted to hospital, and how their treatment needs to be increased or decreased during infection.

The aim is to recruit 100 patients admitted to hospital due to a respiratory infection. It is voluntary to take part and participants can choose to withdraw at any time. The study will involve some blood and nose samples. This will be done on Day 0, Day 2 and Discharge from hospital, and an out-patient follow-up visit on Day 28. The data will be used to develop novel diagnostic tools to assist in rational treatment decisions that will benefit both individual patients and resource allocation. It will also establish research preparedness for upcoming pandemics.

DETAILED DESCRIPTION:
Despite clinical advances and decades of research, the ability to reliably predict the course of respiratory viral diseases such as influenza and coronavirus infections remains poor. The aim of this project is to develop a platform for identifying and developing predictive tests by combining physiological data and correlates of severity in influenza-like infections so that progression to severe pulmonary involvement can be anticipated during respiratory viral infection. This would then permit safe discharge of patients with self-limiting disease or more rapid intensification of treatment as appropriate.

Respiratory infections are among the most important causes of severe disease worldwide, with the major respiratory viruses responsible for overwhelming pressure on health services each winter due to annual surges in incidence. The two most common viral causes of severe lung disease, influenza and respiratory syncytial virus (RSV), are responsible for ~50% of hospital admissions in children and 22% in adults, with mortality greatest in older people. As the population ages, this burden of disease is steadily increasing. Furthermore, the continual risk of newly emergent pandemic influenza strains that arise unpredictably is universally considered one of the most critical threats to global health and socioeconomic stability. This has been demonstrated by the recent COVID-19 pandemic.

Risk factors for severe influenza have been investigated extensively in clinical cohorts, with older age, co-morbidities, obesity and pregnancy all increasing the likelihood of severe disease. However, accurate prognostic markers remain elusive and the dynamics of the response to respiratory viral infection has not been explored in naturally-infected patients. Furthermore, biomarker discovery has been limited by heterogeneity in virus strain and dose; delays in timing of presentation; and patient-level confounders. To address these issues, the investigators have conducted controlled human infections with influenza and RSV since 2010, to investigate mechanisms of immunopathogenesis with a particular focus on disease in the human respiratory tract. Recent preliminary data from a cohort of volunteers infected with the influenza A(H1N1)2009 strain showed that rapid changes in the transcriptome of whole blood occurred within 2 days of virus exposure. During the 2009 influenza pandemic, similar studies were also performed with hospitalised patients. There, transcriptomic analysis of blood showed similar antiviral signatures in less severely unwell individuals but divergent signatures associated with poor clinical outcomes.

The aim of this project is to identify and test predictors of disease progression and clinical deterioration in patients with influenza-like illness, in order to develop novel methods to more accurately determine the need for hospital admission and treatment intensification during respiratory viral infection. To further develop and test these biomarkers in an independent cohort of naturally-infected patients, hospitalised adults with influenza-like illness will be recruited within 24 hours of admission and samples obtained from blood and nose at 3 subsequent time-points.

Using these data, predictive transcriptomic signatures will be identified. Longitudinal samples and clinical data will then be used to test, validate and refine them in affected local populations. These findings will then be translated into novel diagnostic tools and a biobank established for further investigation of the virology and immunopathogenesis of severe respiratory viral infections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons aged ≥ 18, and able to give informed consent
* Patient is admitted to hospital
* Primary reason for hospital admission is clinical suspicion of a new episode of ARI
* Onset of the following symptoms within the last 7 days: i. Sudden onset of self-reported fever OR temperature of ≥ 38°C at presentation AND ii. At least one respiratory symptom (cough, sore throat, runny or congested nose, dyspnoea) AND iii. At least one systemic symptom (headache, muscle ache, sweats or chills or tiredness).

Exclusion Criteria:

* Patient lacks capacity to provide informed consent
* Patient has been transferred from another hospital
* Patient has been previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-patients admitted to hospital with a confirmed or suspected respiratory infection.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The expectation is that after analysis the data from this study will be widely distributed in the medical and scientific community. Facilitated with presentations at local, national and international meetings, the hope is to publish widely in the medical literature. In addition there is an excellent media department at Imperial College that will publicise research that has public interest when it is published. All data will be anonymised and aggregated or pseudonymised; no identifying participant information will be published.
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available approximately 12 months from the last patient's last visit and remain available indefinitely
Access Criteria: According to study protocol

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Persons Aged ≥ 18 Years: Healthy persons aged ≥ 18 years who meet the inclusion/exclusion criteria
Period: Overall Study
Arm/Group | Healthy Persons Aged ≥ 18 Years
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Persons Aged ≥ 18 Years
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 55 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Mixed (White and Asian) | 2
  Race and Ethnicity: Asian or Asian British (Indian) | 3
  Race and Ethnicity: White British | 2
  Race and Ethnicity: White Other | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Describe the Aetiology of Influenza-like Illness in Hospitalised Adults
Description: The identity of pathological organisms associated with influenza-like illness (including respiratory viruses and bacteria) will be obtained from the patient's medical record
Time Frame: Day 0 to Day 28
Population: 8 participants were enrolled into this study with a diagnosis of ARI (Acute Respiratory Infection)
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Persons Aged ≥ 18 Years
Number analyzed (Participants) | 8
Participants
  SARS-CoV-2 | 4
  No pathogen | 4

2. Primary Outcome: Describe the Clinical Outcomes of Influenza-like Illness in Hospitalised Adults
Description: Data collection on Day 28 will consist of clinical diagnosis at discharge, any febrile illness in the 7 days preceding the visit, mortality and complications between Day 0 and 28.
Time Frame: Day 0 to Day 28
Population: 8 participants who were enrolled had a diagnosis of Acute Respiratory Illness (ARI) then recovered and were discharged home.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Persons Aged ≥ 18 Years
Number analyzed (Participants) | 8
Participants
  Acute Lung Injury/Acute Respiratory Distress syndrome | 1
  ARI and hyperglycaemia | 1
  ARI secondary to SARS-CoV-2 infection | 2
  ARI with no causative pathogen found | 1
  ARI with no causative pathogen found with partial middle lobe collapse and anaemia | 2
  ARI with left lower lobe abscess and dermatitis | 1

3. Primary Outcome: Describe the Clinical Management of Influenza-like Illness in Hospitalised Adults
Description: Describe the Clinical Management of Influenza-like Illness in Hospitalised Adults
Time Frame: Day 0 to Day 28
Population: 8 participants were enrolled into this study. 6 participants, 3 of which with confirmed SARS-CoV-2 infection, received a steroid treatment. 7 participants received a treatment course of antibiotics.
  1 participant did not receive any antibiotics, this participant did not have a confirmed causative respiratory pathogen found. 4 participants received Remdesivir (antiviral), three of which had a positive PCR test for SARS-CoV-2, one without.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Persons Aged ≥ 18 Years
Number analyzed (Participants) | 8
Participants
  Antibiotic + Steroid Treatment | 3
  Antibiotic Treatment | 1
  Antibiotic + Antiviral Treatment | 1
  Antibiotic + Antiviral + Steroid Treatment | 2
  Antiviral + Steroid Treatment | 1

4. Secondary Outcome: Identify Changes in Cytokine Levels During Influenza-like Illness in Hospitalised Adults
Description: Cytokine levels (in pg/mL) will be measured in plasma and nasal lining fluid samples by MesoScale Discovery
Time Frame: Day 0 to Day 28
Population: As we only recruited 8 participants out of the 100 recruitment target, the cytokine assays were not run and therefore no results are available for this outcome measure due to the poor recruitment.
Arm/Group | Healthy Persons Aged ≥ 18 Years
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 0 to Discharge or Day 28 (whichever came first)
Description: Adverse Events and Serious Adverse Events were captured from the time of consent until the time of discharge.
Arm/Group | Healthy Persons Aged ≥ 18 Years
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Persons Aged ≥ 18 Years (N=8)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
This study only recruited 8 participants of the 100 total recruitment target.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT04664075/Prot_SAP_000.pdf